CLINICAL TRIAL: NCT00005643
Title: Evaluation of Doxil in the Treatment of Recurrent or Advanced Leiomyosarcoma of the Uterus
Brief Title: Chemotherapy in Treating Patients With Sarcoma of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067809; GOG-0087J
Record Dates: First submitted 2000-05-02; First posted 2004-04-19 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2005-11

CONDITIONS: Endometrial Cancer; Sarcoma
Keywords: stage IV uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Sarcoma; Sarcoma, Endometrial Stromal

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating patients who have advanced or recurrent sarcoma of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of doxorubicin HCl liposome in patients with recurrent or advanced uterine sarcoma. II. Determine the nature and degree of toxicity of this drug in this patient population.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 1 hour. Treatment continues every 4 weeks in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced, persistent or recurrent uterine sarcoma with documented disease progression after appropriate local therapy Leiomyosarcoma Malignant mixed mullerian tumor (mixed mesodermal tumor, mixed heterologous mesenchymal sarcoma) Mixed malignant Muellerian tumor (carcinosarcoma, homologous mesenchymal sarcoma) Endometrial stromal sarcoma Other uterine sarcomas Considered incurable Bidimensionally measurable disease consisting of abdominal, pelvic, chest, or other masses by palpation, x-ray, computed tomography, or ultrasound

PATIENT CHARACTERISTICS: Age: Over 21 Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: LVEF normal by MUGA scan Other: No clinically significant infection No other malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior therapy with cytotoxic drugs No prior doxorubicin HCl liposome No prior doxorubicin greater than 360 mg/m2 No other concurrent antineoplastic agents Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy No prior radiotherapy for any other malignancy Surgery: Recovered from prior surgery Other: No other concurrent investigational agents

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Sutton, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (49):
- United States (48):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Sutton G, Blessing J, Hanjani P, Kramer P; Gynecologic Oncology Group. Phase II evaluation of liposomal doxorubicin (Doxil) in recurrent or advanced leiomyosarcoma of the uterus: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Mar;96(3):749-52. doi: 10.1016/j.ygyno.2004.11.036. PMID 15721421